# **Informed Consent**

Study Title: Akashic Records and Mental Health Outcomes

ClinicalTrials.gov Identifier: NCTXXXXXXX

Document Type: Informed Consent

Revision Date: [5.21.24]

Principal Investigator: Candice S. Rasa, LCSW

Co-Investigator: Sarah Coleman, LCSW

Sponsor: Rasa Healing, Inc.

#### **Informed Consent Form**

Title: How Akashic Records Sessions Affect Mental Health

#### **Principal Investigator and Sponsor**

Candice S. Rasa, LCSW 901 SW Martin Downs Blvd, Suite 303, Palm City, Fl 34990 (954) 610-7961 candice@rasahealingservices.com

## **Independent Evaluator**

Sarah Coleman, LCSW (305) 735-9192 va.research@rasahealingservices.com

#### **Research Coordinator**

Betsy Koczab (561) 316-3414 va.admin@rasahealingservices.com

# **Research Consent Summary**

You are being asked for your consent to take part in a research study. This document provides a summary of this research and expectations for participating. It describes the key information that most people need to decide whether to take part in this research.

#### What should I know about this study?

- Someone will explain this research to you.
- Taking part in this research is voluntary. Whether you take part is up to you.
- If you don't take part, it will not affect your receipt of clinical services.
- You can take part now and later drop out, and it won't be held against you. You will not be billed for canceling an Akashic Record session.
- If you don't understand something, you are encouraged to ask questions.
- You can ask all the questions you want before you decide if you want to participate.

# **Key Information**

You're invited to join a study to see how two Akashic Record sessions might affect how you feel. We're looking at stress, anxiety, depression, resilience, and feeling connected. Rasa Healing is sponsoring this study. We want to know: Can Akashic Records sessions make mental health

better? We'll see if stress, anxiety, and depression go down, and if you feel stronger and more connected to yourself and to others.

There might be some tough moments, like thinking about your life and your feelings. But you might also understand Akashic Records better and learn more about yourself. You'll have two sessions with Candice Rasa, LCSW. Everything you say will stay private.

If you've had an Akashic Record session before with someone else, this might be different. If it's your first time, you might not know much about it. Candice Rasa will answer any questions you have during your first session. This is the first time Akashic Record sessions are being studied in a clinical trial.

If you join this study, you won't be able to have more sessions with Candice Rasa until after the study is done. We also want any therapy you're doing to stay the same while you're in the study.

# What to Expect

Around 100 people will be part of this study. If you agree to participate, this study should take approximately six hours of your time across 3 months and 2 weeks.

This study will use competitive enrollment. This means that once the target number of people begin the study, all further enrollment will be closed. Therefore, it is possible that you may have filled out the pre-screen questionnaire, but not be invited to continue with the study if the target number of people has already been reached. We will let you know when the study is closed for new applicants whenever we make that decision. We reserve the right to close the study at any time.

#### **Study Timeline**

# **Phase 1: Application and Approval Process**

- o Initial Application: 10-20 minutes
- o Pre-screen Interview: Approximately 1 hour
- Read and Sign paperwork: 10 minutes
  - Minimum 1 day prior to the first Akashic session. It must be completed before your session.

#### Phase 2: Self Assessments and Akashic Sessions

- First self-report assessment scales: 15 minutes
  - Within 7 days of the 1st Akashic session. Must be completed before the session.
  - Demographic Form
  - CD-RISC-10 Connor Davidson Resilience Scale
  - DASS-21 Depression and Anxiety Scale
  - Watt's Connectedness Scale
- o Initial Akashic Session: 90 minutes

- No later than 30 days after pre-screen (or additional pre-screen will need to be conducted)
- Second set of self-report assessment scales: 15 minutes
  - Must be completed within 7 days of the second Akashic session. Must be completed prior to starting the second session.
  - CD-RISC-10 Connor Davidson Resilience Scale
  - DASS-21 Depression and Anxiety Scale
  - Watt's Connectedness Scale
- Second Akashic session: 50 minutes
  - 10-21 days after the first session

#### Phase 3: Final Assessments and Semi-Structured Interview

- Third set of self-report assessment scales: 15 minutes
  - 7-14 days after the 2nd Akashic session. Must be completed prior to semi-structured interview.
  - CD-RISC-10 Connor Davidson Resilience Scale
  - DASS-21 Depression and Anxiety Scale
  - Watt's Connectedness Scale
  - Satisfaction Survey
- Potential Semi-Structured interview: Approximately 1 hour
  - 7 to 14 days after the final Akashic session
- Fourth set of self-report assessment scales: 15 minutes
  - 60 to 80 days after final Akashic session
  - CD-RISC-10 Connor Davidson Resilience Scale
  - DASS-21 Depression and Anxiety Scale
  - Watt's Connectedness Scale

# What happens to me if I agree to take part in this research?

If you qualify to take part in this study and go on to receive the study treatment, then the following will happen:

**Self-Report Scales:** Before and after each session, you'll need to fill out forms to show how stressed, anxious, or sad you feel, and how resilient and connected you feel. Everyone will need to complete these assessments for every session, and also fill out a satisfaction survey one time at the end of the study.

| Demographic Survey x1 |
|------------------------------------------------|
| CD-RISC-10 Connor Davidson Resiliency Scale x3 |
| DASS-21 Depression and Anxiety Scale x3 |
| Watt's Connectedness Scale x3 |

| ☐ Satisfaction S | Survey | x1 |
|------------------|--------|----|
|------------------|--------|----|

**Akashic Records Session(s)**: You will take part in two Akashic Records sessions. During these sessions, Candice Rasa, LCSW, will connect to the Akashic Record for you. Candice is both a licensed clinical social worker and a certified Akashic Records channel. This record is like a cosmic library where all information is stored. People who channel the Akashic Record use special senses like intuition to understand and interpret this information, which they then share with you. These sessions usually involve talking about past experiences, emotional patterns, and other personal topics. Candice will provide suggestions and resources fit to your needs.

Each session will last about 50-90 minutes and will be scheduled at times that work for both you and Candice. You'll have the freedom to choose what you talk about during the sessions. You can ask questions and talk about what's important to you. The sessions will be completed using a secure platform called Google Meet. These sessions will be recorded. After each session, the recording will be stored securely online, and you'll have seven days to download it. These recordings might be studied later for more insights, but they won't be shared with anyone outside of the research team.

**Semi-structured Interview:** Some of you may be asked to be interviewed about a week after your last Akashic reading. This interview will allow you to talk in more detail about your experiences. However, not everyone will be chosen for this interview. Our goal is to complete 30 to 50 interviews for this study, but we'll decide when to stop based on what we learn. If you do take part in an interview, it will last about an hour. During the interview, you can talk about what you felt during and after the Akashic Records sessions.

These interviews will be recorded and kept safe using a password protected Google Workspace, which is secure and follows privacy laws. Afterward, the interviews will be written down, and any names or personal details will be removed. Once the study is over, the recordings will be deleted from Google Workspace to ensure your privacy and stored on a secure jump drive for 6 years.

**Risks**: Taking part in this study could have potential risks. These include feeling uncomfortable when filling out forms, answering personal questions during interviews, or thinking deeply about your life and feelings. During the Akashic sessions, you might remember things that upset you or feel strong emotions. Personal growth might happen slowly over time, and you might not feel as spiritually connected as you hoped. There could be other emotional risks we don't know about yet, and you are welcome to stop the session or interview at any time if you feel uncomfortable.

**Benefits**: These sessions could have a positive impact and help you deal with personal problems right away. You might gain a better understanding of your feelings and why you have them. They could help you discover hidden strengths and make you feel stronger and more at peace with yourself.

**Alternatives to Participation:** If you don't want to join the study, but you still want help for your mental health, we will help you. You can get help from a licensed mental health professional. We can refer you to mental health experts in your area.

# What happens to the information collected for this research?

The data collected and saved from this study will be de-identified, meaning that no one will be able to identify you from the data. That information includes your name, initials, or full birth date. Instead, you'll have a special code just for this study. If we publish or talk about the study's results, we won't include your name. The de-identified data might also be used in future studies or by other researchers. We will not ask for your permission again to use this data in future studies.

All the information we gather will be kept private and stored safely. We'll keep records of your involvement in the study confidential, except if we're legally required to share it or as explained in this form. The sponsor and sometimes the Institutional Review Board (IRB), may review and copy study records that have your name. This means we can't promise absolute secrecy, but only authorized research personnel will have access to this data.

- Sarah Coleman, LCSW Co-Investigator, Independent Evaluator
- Candice Rasa, LCSW Akashic Records Channel, Principal Investigator
- Betsy Koczab, VA Research Coordinator
- Briana Williams, Research staff
- Rasa Healing, Inc., Sponsor
- Institutional Review Board

By signing this form, you allow the above people to access your name, your self-assessments, and your interview answers for research purposes. You also agree to let them use your direct quotes in articles, knowing that you will remain anonymous. The research team won't share any info that could identify you.

You won't get individual results from this study, but you can track your own self-assessment scores if you want.

#### **Voluntary Participation and Withdrawal:**

Your participation in this study is voluntary. If you decide not to take part, there will be no penalty or loss of benefits that you are otherwise entitled to. You can also stop participating at any time without any penalty or loss of benefits.

The research team can also end your participation for the following reasons:

- If there's an urgent mental health situation and you need help right away to keep you safe.
- If you're not following the rules or directions of the study.
- If it's found out that you don't meet the requirements for the study.
- If the study itself is stopped for any reason.

If we find out any important new information during the study that might change your mind about staying in the study, we will tell you right away. This includes any new details about the risks, benefits, or anything else that might affect your decision to continue. We want to make sure you have all the information you need to decide if you want to keep being part of the study.

## **Compensation:**

You won't get paid for joining this research. But you will get a 15% discount on each Akashic Record session.

Here's how it works: The first session is 90 minutes and costs \$379 but for research participants it costs \$322. Follow-up sessions typically cost \$239, but you'll only pay \$203.

Overall, you'll save \$93 on both sessions by being part of the study.

You'll get help setting up your sessions to fit the study schedule.

#### **Contact Information:**

For questions or concerns regarding the study, you may contact the following people: Sarah Coleman at <a href="mailto:va.research@rasahealingservices.com">va.research@rasahealingservices.com</a>
Candice Rasa at <a href="mailto:candice@rasahealingservices.com">candice@rasahealingservices.com</a>
Betsy Koczab at <a href="mailto:va.admin@rasahealingservices.com">va.admin@rasahealingservices.com</a>

An institutional review board (IRB) is an independent committee established to help protect the rights of research subjects. If you have any questions about your rights as a research subject, contact (Monday through Friday 9-5 EST/EDT):

By mail: Pearl IRB 29 East McCarty Street Suite 100 Indianapolis, IN 46225 https://www.pearlirb.com/

or call: 317-899-9341 (main) or fax: 317-602-6554 (fax)

or by email: support@pearlirb.com

Please reference the IRB study number when contacting the IRB.

#### **Signature For Consent**

Signing this consent form indicates that you:

- 1. agree to participate in this research study;
- 2. agree to complete all assessments, readings, and interviews as outlined above;
- 3. have read and understand the information in this form, which is written in English;
- 4. have had the information in this form explained to you clearly and have had your questions, answered to your satisfaction;
- 5. have access to a signed and dated copy of this form;
- 6. understand that you can withdraw from this study at any time via written or verbal communication; and
- 7. understand that you will not be reimbursed if you withdraw from this study;
- 8. understand you will not be charged a cancellation fee if you reschedule a session or if you decide to withdraw from the study early.

| agree to be a research participant in this research study: | | |
|---|---|---|
| Research Participant's Signature | <br>Date | Time |
| Research Furticipant's Signature | Buc | Time |
| Print Research Participant's Name | | |
| Researcher Signature | Date | Time |
| Print Researcher's Name | | |